CLINICAL TRIAL: NCT03799081
Title: Use of Fetoscopy in Missed Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-00056-18
Record Dates: First submitted 2018-11-05; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed | interventions — Fetoscopy

STUDY DESIGN:
Intervention Model Description: Women who have undergone a missed abortion in the first trimester who want a surgical treatment option
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fetoscopy in missed abortion (Other): Women who have decided to undergo fetoscopy in missed abortion
  Interventions: Procedure: Fetoscopy

INTERVENTIONS:
Procedure: Fetoscopy — Fetoscopy is a procedure that enables viewing of the fetus through use of a hysteroscope

SUMMARY:
The purpose of this study is to evaluate the use of hysteroscopic embryoscopy or fetoscopy as a powerful diagnostic tool to provide better counseling for couples having experienced pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with missed abortion during the first trimester of pregnancy

Exclusion Criteria:

* Women diagnosed with missed abortion after the first trimester of pregnancy
* Any contraindication for hysteroscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Macroscopic anatomic malformations in missed abortions | Two years
  The number and type of macroscopic anatomic malformations in missed abortions will be determined through visual observation using a fetoscope

SECONDARY OUTCOMES:
Minimize intrauterine adhesions through observation | Two years
  To minimize intrauterine adhesions that might occur after curettage through the ability to visualize the womb and pregnancy site through a hysteroscope before the surgical procedure so that inadvertent intrauterine adhesions are minimized. After one year, if pregnancy is not achieved (due to intrauterine adhesions that cause infertility), a follow-up hysteroscopy will be performed and intrauterine adhesions can be visualized if they have occurred.
Prevention of retained conception products | Two years
  Prevention of retained conception products by hysteroscopy after curettage and visualization and observation of the contents of the womb

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Haimovich, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No